CLINICAL TRIAL: NCT05013502
Title: Management of Diuretic Refractory Ascites in Cirrhosis With Empagliflozin (DRAin-Em-01)
Brief Title: Empagliflozin in Diuretic Refractory Ascites
Acronym: DRAin-Em 01
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Aparna Goel, Protocol Director, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-61538
Record Dates: First submitted 2021-08-06; First posted 2021-08-19 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Liver Cirrhosis; Cirrhosis; Ascites; Ascites Hepatic; Sodium-Glucose Transporter 2 Inhibitors
Keywords: diuretic refractory; diuretic resistant; empagliflozin
MeSH Terms: conditions — Liver Cirrhosis; Fibrosis; Ascites | interventions — empagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Empagliflozin 10mg PO daily for 12 weeks (Experimental): Single arm trial
  Interventions: Drug: Empagliflozin 10 MG

INTERVENTIONS:
Drug: Empagliflozin 10 MG — empagliflozin 10mg PO once daily

SUMMARY:
Ascites is the most frequent complication of liver cirrhosis and results in increased morbidity and mortality but current medical management options are limited. Here, the investigators will conduct an interventional single-arm pilot clinical trial toevaluate the feasibility of empagliflozin in managing diuretic-resistant ascites in patients with decompensated cirrhosis. This single site, open label pilot study will enroll participants with decompensated cirrhosis at a single site. Participants will receive empagliflozin 10mg oral tablets once daily for 12 weeks with monitoring for safety and adverse events.

DETAILED DESCRIPTION:
Pharmacologic options for the management of ascites are limited to diuretics only. Each year approximately 10% of patients with cirrhosis develop diuretic-resistant ascites, necessitating the use of more invasive procedures such a paracentesis, transjugular intrahepatic portosystemic shunting (TIPS), and transplantation; each modality is associated with significant risks and limitations. Patients treated with diuretics may also develop complications such as acute kidney injury, encephalopathy, muscle cramping, or hyponatremia, limiting optimal dosages of these medications and hence, resulting in inadequate control of fluid retention. Thus, ascites that is resistant to our current therapies is an important unmet medical need.

Recently, SGLT2-Is have been shown to reduce heart failure hospitalizations and cardiovascular death in patients with and without diabetes in landmark, large-scale clinical trials. Empagliflozin improved heart failure outcomes without altering hemoglobin A1c or increasing risk of hypoglycemia in individuals without diabetes, suggesting that SGLT2-Is may act through a neurohormonal mechanism independent of blood glucose changes. Because cirrhosis and heart failure are disorders with a common pathophysiology of decreased effective arterial blood volume with resultant stimulation of the renin-angiotensin-aldosterone system (RAAS), sympathetic nervous system, and total body fluid overload, the investigators hypothesize that SGLT2-Is may be effective in the management of ascites. Multiple lines of evidence suggest SGLT2-Is may have a beneficial role in chronic liver disease. Several case reports of patients with cirrhosis and diuretic-resistant ascites have found that SGLT2-I treatment was associated with near resolution of ascites and pedal edema. SGLT2-I treatment has also demonstrated improved hepatic function, reduction of fibrosis and normalization of liver enzymes in non-alcoholic fatty liver disease (NAFLD).Although SGLT2-I are partially cleared by the liver, empagliflozin is well tolerated in patients with cirrhosis. Thus, the investigators initiated a feasibility study to test the hypothesis that the SGLT2-I, empagliflozin, will decrease ascites by attenuating maladaptive neurohormonal and inflammatory responses in cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Decompensated liver cirrhosis with ascites
* Diuretic-resistant ascites defined as one of the following: a) An inability to mobilize ascites despite adherence to dietary sodium restriction (2000 mg per day) and administration of maximum tolerable doses of oral diuretics; b) Rapid reaccumulation of fluid after therapeutic paracentesis despite adherence to a sodium-restricted diet. c) Development of diuretic-related complications such as progressive azotemia, hepatic encephalopathy, or progressive electrolyte imbalances
* Ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

* Hypersensitivity to any SGLT2 inhibitor
* Pregnant or breastfeeding women
* eGFR below 45mL/min/1.73m2 or decrease in eGFR by >30% between screening
* Recurrent urinary tract infections or recurrent genitourinary fungal infections, defined as > 2 infections in six months or >3 infections in one year
* Hypotension requiring oral vasopressor therapy
* Patients with particular risk for ketoacidosis including active moderate or severe alcohol use disorder, pancreatitis, pancreatic insulin deficiency from any cause, or episode of ketoacidosis in the past
* History of skin or soft tissue infection requiring IV antibiotics including Fornier's gangrene or prior limb amputation
* Chronic alcohol or drug abuse or any condition that, in the investigator's opinion, makes them an unreliable trial subject or unlikely to complete the trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Participant retention rate as a measure of study feasibility | Baseline to 12 weeks
  Retention rate and completion of trial activities through 12 weeks

SECONDARY OUTCOMES:
Mean change in abdominal girth from baseline to 12 weeks | Baseline to 12 weeks
  Abdominal girth as a measure of ascites volume
Mean change in body weight from baseline to 12 weeks | Baseline to 12 weeks
  Body weight as a measure of ascites volume
Mean change in patient reported functional status | Baseline to 12 weeks
  Functional status and quality of life measured on SF-36 questionnaire
Estimated glomerular filtration rate as a measure of kidney function | Baseline to 12 weeks
  Change in renal function as measured by serum creatinine

CONTACTS AND LOCATIONS:
Overall Officials: Aparna Goel, MD, Principal Investigator — Clinical Assistant Professor
Locations (1):
- Stanford University Digestive Health Clinic, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No